CLINICAL TRIAL: NCT07054320
Title: Rapamycin Treatment for Prevention of Infection-related Illness
Brief Title: Rapamycin and Infection-related Illness
Status: Recruiting | Type: Observational
Sponsor: Hoskinson Health and Wellness Clinic (Industry)
Responsible Party: Principal Investigator, William Hoskinson, Chief Medical Officer, Hoskinson Health and Wellness Clinic
Other Study IDs: BRANY IRB File # 25-02-270-149
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Infectious Diseases
Keywords: Infectious Disease; Infection-related illness; Rapamycin; Rapamune; Sirolimus
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Observational procedures — Patients at the Hoskinson Health and Wellness Clinic qualifying for treatment with Rapamune (Sirolimus) receive a prescription from their physician during clinic visits as part of their standard health care. This study will evaluate the safety, monitor the adverse reactions and observe the preliminary effectiveness of physician-prescribed medical treatment with oral rapamycin [Rapamune (Sirolimus)] in a total of 15 adults, 18 years and older toward preventing and lowering the severity of infectious disease or infection-related illness.

SUMMARY:
Conduct a 6-month observational pilot clinical trial to evaluate the safety, monitor the adverse reactions and observe the preliminary effectiveness of medical treatment with oral rapamycin [Rapamune (Sirolimus)] in a total of 15 adults, 18 years and older toward preventing and lowering the severity of infectious disease or infection-related illness.

Rapamune (Sirolimus) is not approved by the United States Food and Drug Administration (FDA) to prevent and lessen the severity of infection-related illness or infectious disease. Rapamune (Sirolimus) is approved by the FDA for other indications.

The main procedures in the study include:

* Blood tests to examine cholesterol, lipids, blood platelet counts, inflammation and infection-related health parameters
* Questionnaires to examine brain function, mental health, symptoms, overall health status and quality of life
* Electrocardiogram (ECG to measure heart function)
* Resting diastolic and systolic blood pressure

DETAILED DESCRIPTION:
There is limited clinical research to support the efficacy of rapamycin toward preventing the incidence and reducing the severity of infectious disease or infection-related illness in humans. The off-label use of rapamycin to prevent infection may be implemented safely in healthy individuals with well-controlled medical conditions and/or prescribed medications compatible with its established indications detailed in the FDA-approved prescription label/medical guide. Pregnant women, organ transplant recipients (especially lung and liver), and patients with cancer, serious wounds or infections, allergies to rapamycin and its derivatives, hyperlipidemia and recent vaccinations are particularly compromised. Short term dosing regimens are generally well-tolerated with mild to moderate adverse events and no severe adverse events in patients qualifying and receiving treatment. Long term use should be evaluated further, and the use of rapamycin derivatives in healthy patients as an infection preventive therapy warrants further investigation.

This study proposes to observe the following parameters prior to, and at 3 and 6 months after the initiation of the observational study:

* Safety [no. and level of adverse events, MSQ, SPB and DPB, blood platelet counts, lipid profiles, ECG, cognitive function, depression symptoms, systemic inflammation, urinalysis (only in female participants of child-bearing age for pregnancy test)]
* Incidence of infectious disease or infection-related illness
* Severity of infectious disease or infection-related illness
* Incidence of infection-related hospitalizations
* Quality of Life (RAND SF-36 Health Survey)
* Global Health Questionnaire (PROMIS-GHF V1.2)
* Patient Self-Report Questionnaire of symptoms, incidence and severity of infectious disease or infection-related illness and hospitalizations one year prior and 3 and 6 months following the initiation of the observational study.

Patients at the Hoskinson Health and Wellness Clinic qualifying for treatment with (Rapamune (Sirolimus) receive a prescription from their physician during clinic visits as part of their standard health care. Patients do not have to participate in this study to receive medical treatment with Rapamune (Sirolimus) for their condition.

Measurement of infection related illness parameters [Complete Blood Count (CBC), White Blood Cell Count (WBC), Neutrophils, Lymphocytes, Eosinophils, Basophils, Monocytes, C-Reactive Protein (CRP), Procalcitonin (PCT), Erythrocyte Sedimentation Rate (ESR), Absolute Neutrophil Count (ANC)], fasting total cholesterol (TC), High (HDL) and Low (LDL) lipoproteins and triglycerides, inflammatory biomarkers (CRP, Tumor Necrosis Factor (TNFα), requires a blood draw, which is associated with some discomfort and minor risks such as a slight bruising of the arm. A registered nurse will be available to assist with all blood draws/testing. Study participants will be advised of the known risks and consequences associated with the testing and also of the reasonably known risks and consequences of not undergoing testing.

The Quality of Life (RAND SF-36 Health Survey), Global Health Questionnaire (PROMIS-GHF V1.2) Patient self-report questionnaire, systolic blood pressure (SPB) and diastolic blood pressure (DPB), electrocardiogram (ECG), medical symptoms questionnaire (MSQ), Cognitive function by Montreal Cognitive Assessment [MoCA (Jak-Bondi Criteria)] and Advanced Digital Cognitive Assessment (BrainCheck)], Depression by the Center for Epidemiologic Studies Depression Scale (CES-D Scale) are non-invasive and no adverse reactions or side effects are expected.

As with any routine clinical care paradigm, other primary potential risks include a breach of confidentiality and loss of privacy from unauthorized disclosure of the study participants' personal health information. Such events could conceivably lead to economic loss for patients through discriminatory practices. However, this study presents minimal risks to the study participants whose data are being analyzed because rigorous precautions will be employed to protect privacy, confidentiality and security of personal health information. These precautions are outlined in the Data and Safety Monitoring Plan (DSMP).

Study participants will be advised of the known risks and consequences associated with the testing and also of the reasonably known risks and consequences of not undergoing testing. A physician will be present at each testing visit to assess any potential side effects or complications. A registered nurse will be in attendance to assist with all testing. The investigators are experienced in providing a safe environment where study participants feel comfortable, especially with tests that require them to remain motionless for extended periods of fame.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female Adults, 18 years and older
* Females of child-bearing age taking birth control medication
* Received a Hoskinson Health and Wellness Clinic physician prescription for Rapamune (Sirolimus)

Exclusion Criteria:

* Adults requiring monoclonal antibody or biological treatment
* Adults diagnosed with an acute lower respiratory or GI infection within 2 weeks
* Adults females who are not taking birth control medication, are pregnant or nursing mothers
* Adults reporting severe mental or physical disability
* Adults reporting unwillingness to travel to onsite clinical facilities
* Adults with any change in chronic disease symptoms or medication within 3 months
* Any contraindications to medical treatment with Rapamune (Sirolimus), as outlined in the FDA-approved medication guide

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female adults, 18 years and older
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of infectious disease or infection-related illness | Prior to and 3 and 6 months following the initiation of the observational study
  The Primary Endpoint is the incidence and severity of infectious disease or infection-related illness prior to and 3 and 6 months following the initiation of the observational study measured by:
  * CBC
  * WBC
  * Neutrophils
  * Lymphocytes
  * Eosinophils
  * Basophils
  * Monocytes
  * CRP
  * PCT
  * ESR
  * ANC
  * Incidence of infection-related hospitalizations

SECONDARY OUTCOMES:
Quality of Life (RAND SF-36 Health Survey) | Prior to and 3 and 6 months following the initiation of the observational study
  The RAND 36-Item Health Survey taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. All items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. Items in the same scale are averaged together to create the 8 scale scores.
Global Health Questionnaire (PROMIS-GHF V1.2) | Prior to and 3 and 6 months following the initiation of the observational study
  PROMIS adult Global scale v1.2 produce two scores: Global Mental Health and Global Physical Health. Most questions have five response options ranging in value from one to five. The total raw score for a scale is summed from the appropriate values of the responses from relevant questions. The sum of raw scores is converted into a T-score for each participant. The T-score rescales the raw sum score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean.
Patient self-report questionnaire | One year prior and 3 and 6 months following the initiation of the observational study
  Patient self-report questionnaire of the following outcomes (during the one year prior and 3 and 6 months following the initiation of the observational study):
  * Symptoms of infectious disease or infection-related illness
  * Incidence and severity of physician diagnosed infectious disease or infection-related illness
  * Incidence of infection-related hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: William Hoskinson, DO, Principal Investigator — Hoskinson Health and Wellness Clinic
Locations (1):
- Hoskinson Health and Wellness Clinic, Gillette, Wyoming, United States

IPD SHARING:
Plan to Share IPD: Yes
Study outcome data will be shared upon request to the principal investigator.

REFERENCES:
- [Background] Hays RD, Spritzer KL, Fries JF, Krishnan E. Responsiveness and minimally important difference for the patient-reported outcomes measurement information system (PROMIS) 20-item physical functioning short form in a prospective observational study of rheumatoid arthritis. Ann Rheum Dis. 2015 Jan;74(1):104-7. doi: 10.1136/annrheumdis-2013-204053. Epub 2013 Oct 4. PMID 24095937
- [Background] Rothrock NE, Amtmann D, Cook KF. Development and validation of an interpretive guide for PROMIS scores. J Patient Rep Outcomes. 2020 Feb 28;4(1):16. doi: 10.1186/s41687-020-0181-7. PMID 32112189
- [Background] Wu Q, Chen Y, Zhou Y, Zhang X, Huang Y, Liu R. Reliability, validity, and sensitivity of short-form 36 health survey (SF-36) in patients with sick sinus syndrome. Medicine (Baltimore). 2023 Jun 16;102(24):e33979. doi: 10.1097/MD.0000000000033979. PMID 37327281
- [Background] Gandek B, Sinclair SJ, Kosinski M, Ware JE Jr. Psychometric evaluation of the SF-36 health survey in Medicare managed care. Health Care Financ Rev. 2004 Summer;25(4):5-25. PMID 15493441
- [Background] Brazier JE, Harper R, Jones NM, O'Cathain A, Thomas KJ, Usherwood T, Westlake L. Validating the SF-36 health survey questionnaire: new outcome measure for primary care. BMJ. 1992 Jul 18;305(6846):160-4. doi: 10.1136/bmj.305.6846.160. PMID 1285753
- [Background] Kaeberlein TL, Green AS, Haddad G, Hudson J, Isman A, Nyquist A, Rosen BS, Suh Y, Zalzala S, Zhang X, Blagosklonny MV, An JY, Kaeberlein M. Evaluation of off-label rapamycin use to promote healthspan in 333 adults. Geroscience. 2023 Oct;45(5):2757-2768. doi: 10.1007/s11357-023-00818-1. Epub 2023 May 16. PMID 37191826